CLINICAL TRIAL: NCT00978640
Title: Sirtuin Mediated Effects of 36 h Fast and 1 h Exercise
Brief Title: Sirtuin Mediated Effects of 36 Hour Fast and 1 Hour Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 07.09.2009
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Sirt1 activity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fasting and exercise (Experimental): 36 h fast and 1 h ergometer cycling 50% VO2max
  Interventions: Other: fast and exercise
- exercise (Experimental): 1 h ergometer cycling 50% VO2max
  Interventions: Other: exercise

INTERVENTIONS:
Other: fast and exercise — fasting 36 h and exercise 1 h 50% VO2max
  Arms: fasting and exercise
Other: exercise — exercise 1 h 50% VO2max
  Arms: exercise

SUMMARY:
Hypothesis: during fasting and exercise will there be an activation of sirtuins (Sirt1).

Primarily the investigators will investigate Sirt1 activity in muscle- and fat-biopsies after fasting for 36 hours and after 1 hour of ergometer-cycling at 50 Vo2max.

In addition to this the investigators will investigate the effect of fasting and exercise on the velocity of carbamide synthesis, aminoacid rate of turnover and glucose rate of turnover.

ELIGIBILITY:
Inclusion Criteria:

* healthy men
* Body mass index (BMI) 20-26
* age 18-45 years

Exclusion Criteria:

* any kind of disease
* any use of medicine

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Sirt1 activity | 60 min

SECONDARY OUTCOMES:
secondary will we investigate the effect of fasting and exercise on the velocity of carbamide synthesis, aminoacid rate of turnover and glucose rate of turnover. | 4 h

CONTACTS AND LOCATIONS:
Locations (1):
- mikkel Holm Vendelbo, Aarhus, Jylland, Denmark